CLINICAL TRIAL: NCT03136731
Title: Improving Case-finding Strategies for Celiac Disease in Family Members: a Follow-up Study
Brief Title: Evidence-based Screening Strategies for Celiac Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Katri Kaukinen (Other)
Responsible Party: Sponsor-Investigator, Katri Kaukinen, Professor, MD PhD, Tampere University Hospital
Organization: Tampere University Hospital (Other)
Other Study IDs: Celiac2017
Record Dates: First submitted 2017-03-30; First posted 2017-05-02 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Celiac Disease
Keywords: Celiac disease, Gluten, Microbiome, Genetic
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy family members of celiac disease: Celiac disease screening, no intervention.
  Interventions: Diagnostic Test: Celiac disease antibody screening
- Celiac disease index cases: Assessment of disease related factors, no intervention.

INTERVENTIONS:
Diagnostic Test: Celiac disease antibody screening — Observational parameters
  Groups: Healthy family members of celiac disease

SUMMARY:
Main aim: To find evidence-based screening strategies for celiac disease in high risk groups and to find new biomarkers or biomarker combinations for celiac disease diagnostics and follow-up.

DETAILED DESCRIPTION:
The current project will result in the identification of genetic, environmental or downstream biomedical markers that predict the development of celiac disease at the individual level. Moreover, the markers can be exploited in prediction of specific disease risks, manifestations, comorbidities and complications.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Family member of celiac disease patient
* Cohort 2: Previously diagnosed celiac disease

Exclusion Criteria:

* Cohort 1: No previous celiac disease
* Cohort 2: Celiac disease diagnosis not confirmed

Ages: 6 Months to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteers; cohort 1, 3217 genetically predisposed healthy family members of celiac disease patients (high risk group for celiac disease), Cohort 2, 200 new celiac disease index cases will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 3517 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Forthcoming celiac disease diagnosed by current diagnostic criteria | With in 10 years
  Assessed by positive transglutaminase antibodies, small bowel mucosal villous atrophy

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital / Tampere University, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paavola S, Kurppa K, Huhtala H, Saavalainen P, Lindfors K, Kaukinen K. Coeliac disease re-screening among once seronegative at-risk relatives: A long-term follow-up study. United European Gastroenterol J. 2022 Jul;10(6):585-593. doi: 10.1002/ueg2.12255. Epub 2022 May 25. PMID 35611878
- [Derived] Paavola S, Lindfors K, Kivela L, Cerqueira J, Huhtala H, Saavalainen P, Tauschi R, Kaukinen K, Kurppa K. Presence of high-risk HLA genotype is the most important individual risk factor for coeliac disease among at-risk relatives. Aliment Pharmacol Ther. 2021 Sep;54(6):805-813. doi: 10.1111/apt.16534. Epub 2021 Jul 18. PMID 34278595